CLINICAL TRIAL: NCT00296712
Title: Combined Escitalopram/Bupropion as First Line Treatment for Depression, a Replication.
Brief Title: Are Two Antidepressants a Good Initial Treatment for Depression?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #4653
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Major Depression; Dysthymia; Depression NOS
Keywords: Major Depression; Dysthymia; Depression NOS; Escitalopram; Bupropion; Dual Therapy; Combination Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression | interventions — Escitalopram; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- escitalopram + bupropion (Experimental): patients begin on escitalopram 10 mg/d, then bupropion 150 mg/d is added and each is alternately increased as tolerated to maximal dose of escitalopram of 40 mg/d and of bupropion of 450 mg/d
  Interventions: Drug: escitalopram + bupropion

INTERVENTIONS:
Drug: escitalopram + bupropion — same dosing as for monotherapy arms
  Other Names: escitalopram = Lexapro; bupropion = Wellbutrin

SUMMARY:
Relatively drug naive patients will receive two antidepressant medications as initial treatment.

DETAILED DESCRIPTION:
While antidepressant medications are often effective in relieving depressive symptoms, at least 60% of patients do not remit with the first agent tried. This pilot study will assess whether giving two standard medications simultaneously (i.e., Escitalopram and Bupropion) is both tolerated and improves response while decreasing drop outs. This is a replication of a previous study.

ELIGIBILITY:
Inclusion Criteria:

* Currently depressed (DSM-IV Major Depression, Dysthymia or Depression NOS)
* HAMD-D (21-Item) > 9

Exclusion Criteria:

* Prior ineffective adequate trial on either study medication ($ 4 weeks on either escitalopram >20 mg/d or bupropion >300 mg/d; >4 weeks on citalopram >40 mg/d)
* History suggesting increased risk for Seizures (e.g., prior Seizure as an adult, diagnosed Seizure Disorder, taking medication known to increase seizure risk, history of significant head trauma, history of Bulimia or Anorexia)
* History of intolerance to either study medication unless patient and M.D. agree side effect is probably manageable
* Alcohol and/or drug abuse/dependence during past year
* Major medical problems that are not well controlled (e.g., untreated hypertension or diabetes)
* Bipolar I, Bipolar II
* History of Psychosis, or current Psychosis
* Currently taking antidepressants or mood stabilizers, which is judged unwise to discontinue (occasional sleep medication or benzodiazepine for Anxiety is allowed)
* Not currently depressed (whether considered due to current treatment or not)
* Active suicidal risk (history of suicide attempts will be evaluated on a case by case basis)
* Pregnant or breast-feeding
* Premenopausal women not using known effective birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale (HAM-D) | 10 weeks

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI) | 10 weeks
Clinical Global Impression Scale (CGI) | 10 weeks
Patient Global Impression Scale (PGI) | 10 weeks
Arizona Sexual Experience Scale (ASEX) | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Stewart, MD., Principal Investigator — New York State Psychiatric Institute - Columbia University Department of Psychiatry
Locations (1):
- Depression Evaluation Service - New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Stewart JW, McGrath PJ, Deliyannides RA, Quitkin FM. Does dual antidepressant therapy as initial treatment hasten and increase remission from depression? J Psychiatr Pract. 2009 Sep;15(5):337-45. doi: 10.1097/01.pra.0000361276.88339.44. PMID 19820552
- See also: Depression Evaluation Service - official website — http://www.depression-nyc.org
- See also: New York State Psychiatric Institute - official website — http://www.nyspi.org